CLINICAL TRIAL: NCT04425798
Title: Connectivity Alterations of Brain Network in LGG Patients After Levetiracetam Application at Short Term
Brief Title: Connectivity Alterations After Levetiracetam Application
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Beijing Neurosurgical Institute (Other)
Collaborators: Beijing Tiantan Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: KY 2019-038-03
Record Dates: First submitted 2020-06-02; First posted 2020-06-11 (Actual); Last update posted 2020-06-11 (Actual); Status verified 2020-05

CONDITIONS: Glioma; Epilepsy
Keywords: glioma; glioma-related epilepsy; levetiracetam; connectivity alteration
MeSH Terms: conditions — Glioma; Epilepsy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with LEV application: LGG patients with GRE take levetiracetam less than 1 month preoperatively. These patients take levetiracetam tablets twice a day, and one tablet at a time. Each levetiracetam tablet contains 500mg levetiracetam.
- Patients without LEV application: LGG patients with GRE do not take any medicine or receive any treatment preoperatively.

SUMMARY:
This study aimed to analyze the connectivity alterations in brain networks of LGG patients with epilepsy who take levetiracetam at short-term preoperatively.

DETAILED DESCRIPTION:
Glioma-related epilepsy (GRE) is a very common symptom in patients with diffuse gliomas. Approximately 60% of patients with low-grade gliomas (LGGs) and 40-64% of patients with high-grade gliomas presented with GRE at the onset. Although beneficial for the control of GRE, the overall therapeutic effect was unsatisfied and over 20% of patients still suffered from seizures.

GRE was found to be associated with brain network and functional connectivity. And it has been reported that temporal lobe seizures could induce functional connectivity and decreased network efficiency of brain networks. However, the alterations in functional networks induced by GRE were still unclear. And LGG patients with GRE usually take levetiracetam (LEV) preoperatively, which could effectively reduce abnormal spike activity and further cause connectivity alterations. This makes it more complex to reveal the connectivity alterations of brain networks in LGG patients with GRE.

This study aimed to collect the resting-state functional MRIs of 30 LGG patients who presented with GRE at the onset. Through further applied graph theory analysis, investigators tend to reveal the connectivity alterations of brain networks caused by levetiracetam. The findings of this study will provide a theoretical basis for further study of connectivity alterations of brain networks in patients with GRE.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years;
* Histopathological diagnosis with LGG according to the 2016 World Health Organization (WHO) criteria;
* Participants received more than 6 years of school education;
* Presence of GRE, take levetiracetam less than 1 month; or do not take any medicine and receive any treatment;
* No history of biopsy, radiotherapy, or chemotherapy.

Exclusion Criteria:

* Contraindications for MRI;
* Head motion greater than 3 mm in translation or 3° in rotation;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients with LGG presented GRE, take levetiracetam less than 1 month; or do not take any medicine and receive any treatment.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2022-05-25 (Estimated); Primary Completion 2022-05-31 (Estimated); Study Completion 2022-09-30 (Estimated)

PRIMARY OUTCOMES:
The connectivity alterations of brain networks in patients with and without levetiracetam application | through study completion, an average of 2 years
  Graph theory analysis is used to delineate topological networks with resting-state functional MRIs and investigated the characteristics of functional networks. Global and nodal topological properties of brain networks are calculated in the two groups of patients. The difference of topological properties of brain networks between patients with and without levetiracetam application are analyzed using t-test or chi-square test according to the type of data.

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Neurosurgical Institute and Beijing Tiantan Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No
We do not plan to share individual participant data with other researchers